CLINICAL TRIAL: NCT02728167
Title: Randomized, Open-label, Phase II Study to Evaluate the Efficacy of High-Intensity Focused Ultrasound Assisted Hepatic Resection (HIFU-AR) on Blood Loss Reduction in Patients With Liver Metastases Requiring Hepatectomy
Brief Title: Efficacy of HIFU-AR on Blood Loss Reduction in Patients With Liver Metastases Requiring Hepatectomy
Acronym: HIFU-AR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIFU-AR
Record Dates: First submitted 2016-03-22; First posted 2016-04-05 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Liver Metastasis
Keywords: Hepatectomy; Liver metastasis; High-Intensity Focused Ultrasound; Liver metastases (LM) requiring surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-coagulation by HIFU-AR (Experimental): Pre-coagulation of the liver parenchyma with HIFU and standard liver resection
  Interventions: Device: Pre-coagulation of the liver parenchyma with HIFU
- Standard liver resection (No Intervention): Standard liver resection

INTERVENTIONS:
Device: Pre-coagulation of the liver parenchyma with HIFU — 6 to 10 (or more if necessary) side-to-side 40-seconde HIFU treatments
  Arms: Pre-coagulation by HIFU-AR

SUMMARY:
The purpose of this study is to evaluate whether HIFU-assisted liver resection (HIFU-AR) results in reduced blood loss compared to standard liver resection in patients with LM.This is a prospective, monocentric, randomized (1:1 ratio), comparative, open-label Phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the day of consenting to the study.
* Patients with liver metastases requiring a hepatectomy for ≥ 2 segments.
* ECOG PS ≤ 1.
* Adequate bone marrow and liver function at baseline as defined below:

  * Platelet count ≥ 100 x 109/l, and hemoglobin of ≥ 9 g/dl),
  * Total bilirubin ≤ 1.5 x ULN, AST and ALT ≤ 5 x ULN.
* Recovered from prior anti-neoplasic treatment-related toxicity (grade <2 persistent treatment-related toxicity as per CTCAE v4 are accepted).
* Willingness for follow-up visits.
* Covered by a medical insurance.
* Signed and dated informed consent document indicating that the patient has been informed of all aspects of the trial prior to enrolment.

Exclusion Criteria:

* Patients having previously undergone

  * a major hepatic surgery (i.e. more than 3 liver segments) or
  * biliary major surgery.
* Patient with cirrhosis or sinusoidal obstruction syndrome with portal hypertension.
* Pregnant women (women of childbearing potential are required to have a negative pregnancy test within 72 hours prior to inclusion). A positive urine test must be confirmed by a serum pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Normalized blood loss (ml/cm2) | During hepatectomy
  To compare the blood loss during hepactectomy in patients treated by HIFU-AR versus standard liver resection

SECONDARY OUTCOMES:
Total blood los (ml) | During hepatectomy
Transection time | During hepatectomy
Transection time/cm2 of liver area (min/cm2) | During hepatectomy
Hemostasis time | During hepatectomy
Clip density on the liver section area | During hepatectomy
  Number of clips/cm2
Rate of Pringle manoeuvre | During hepatectomy
Rate of patients needing a blood transfusion | During hepatectomy
Length of hospital stay | 10 days
Number of patients with postoperative complications assessed using Dindo-Clavien classification | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michel RIVOIRE, MD, PhD, Principal Investigator — Centre Leon Bérard
Locations (1):
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dupre A, Perol D, Blanc E, Peyrat P, Basso V, Chen Y, Vincenot J, Kocot A, Melodelima D, Rivoire M. Efficacy of high-intensity focused ultrasound-assisted hepatic resection (HIFU-AR) on blood loss reduction in patients with liver metastases requiring hepatectomy: study protocol for a randomized controlled trial. Trials. 2017 Feb 6;18(1):57. doi: 10.1186/s13063-017-1801-2. PMID 28166812